CLINICAL TRIAL: NCT01606553
Title: The INCA Study: Inspiratory Muscle Training in Patients With Chronic Heart Failure
Brief Title: Inspiratory Muscle Training in Patients With Chronic Heart Failure
Acronym: INCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCA
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; respiratory muscle weakness; inspiratory muscle training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-intensity IMT (Experimental): High intensity short duration respiratory muscle training (IMT) using a dual-vave prototype
  Interventions: Device: High-intensity IMT
- Sham High-intensity IMT (Active Comparator): High intensity short duration respiratory muscle training (IMT) using a sham dual-vave prototype
  Interventions: Device: Sham High-intensity IMT

INTERVENTIONS:
Device: High-intensity IMT — High intensity short duration respiratory muscle training with a valve prototype
  Other Names: Orygen-Dual valve prototype
  Arms: High-intensity IMT
Device: Sham High-intensity IMT — High intensity short duration respiratory muscle training using a sham valve prototype
  Other Names: Sham Orygen-Dual valve prototype
  Arms: Sham High-intensity IMT

SUMMARY:
The purpose of this study is to determine whether a high intensity short duration inspiratory muscle training is feasible, secure and effective to improve respiratory muscle function (strength and resistance), health-related quality of life, and to assess potential correlations with health resources utilization.

DETAILED DESCRIPTION:
Patients with chronic heart failure (CHF) often refer exercise intolerance, marked fatigue and dyspnea at low exercise intensities. This characteristic feature might be generated by respiratory and skeletal muscle dysfunction, and it´s has been described as a comorbid status, reflecting the systemic impact of heart failure. Despite the availability of effective pharmacologic treatments, patients with CHF continue to experience progressively worsening symptoms, frequent hospital admission and premature death. Reduced physical functioning, role limitation, and lack of energy may interfere with daily activities as the condition worsens and thereby severely reduce the quality of life in CHF patients. The ACCF/AHA Guidelines for the diagnosis and management of heart failure recommend exercise training as an adjunctive approach to improve clinical status in stable adult patients with current or prior symptoms of heart failure and reduced left ventricular ejection fraction. A wide variety of studies have focussed on respiratory muscles abnormalities in CHF patients. Reduced strength and endurance of respiratory muscles are currently recognized as additional factors implicated in the limited exercise response and quality of life, as well as in a poor prognosis. Additionally, inspiratory muscle training (IMT) has shown to result in improvements on inspiratory strength, functional capacity, ventilatory response to exercise, recovery oxygen uptake kinetics, and quality of life of CHF patients with respiratory muscle weakness. The optimal training scheme remains still to be defined. Most of clinical trials have demonstrated the effectiveness of a low-intensity IMT (maximum 38 cmH2O), but there is little information of the training effects when using higher training loads. Our research group has demonstrated that a short-time high-intensity respiratory training in patients with chronic obstructive pulmonary disease afford to reach good functional results in a shorter time, which affords to make more efficient in terms of time the rehabilitation program and to reach to more patients.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years;
2. chronic heart failure (CHF) of any etiology;
3. clinically stable condition, with no worsening of heart failure or change in cardiac medication in the previous 3 months and during the study; and
4. ability to understand and accept the trial procedures and to sign an informed consent form in accordance with national legislation.

Exclusion Criteria:

1. previous history of any chronic respiratory disease;
2. not to have performed any kind of general or respiratory training in the previous 3 months.

   * Prior to randomization, all patients' clinical assessment and echocardiographic measurements were done by a cardiologist and all patients underwent pulmonary function tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in respiratory muscle function strength | Baseline to 4 weeks
  Transducer measuring maximal inspiratory and expiratory pressures

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline to 4 weeks
  Minnesotta Living wih Heart Failure Questionnaire and Short Form 36
Adverse effects from training | Baseline to week 4
  Adverse events collection by investigator
Health care utilization | Baseline to one year
  Hospital admissions and emergency room visits

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Escalada, MD, PhD, Study Director — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Marco E, Ramirez-Sarmiento AL, Coloma A, Sartor M, Comin-Colet J, Vila J, Enjuanes C, Bruguera J, Escalada F, Gea J, Orozco-Levi M. High-intensity vs. sham inspiratory muscle training in patients with chronic heart failure: a prospective randomized trial. Eur J Heart Fail. 2013 Aug;15(8):892-901. doi: 10.1093/eurjhf/hft035. Epub 2013 Mar 19. PMID 23512093